CLINICAL TRIAL: NCT02359370
Title: The Effects of Lidocaine and Magnesium Sulphate on the Attenuation of the Hemodynamic Response to Tracheal Intubation: Single Center, Prospective, Double-Blind and Randomized Study
Brief Title: The Effects of Lidocaine and Magnesium Sulphate on the Attenuation of the Hemodynamic Response to Tracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, TSA, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LidovsMgOTI
Record Dates: First submitted 2015-01-31; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Intubation Complication; Cardiovascular Morbidity
Keywords: Laryngoscopy; Tracheal Intubation; Lidocaine; Magnesium Sulphate; Cardiovascular Physiological Phenomena
MeSH Terms: interventions — Lidocaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium Group (Active Comparator): Magnesium Sulphate was administered through continuous infusion, immediately before induction of anesthesia
  Interventions: Drug: Magnesium Sulphate
- Lidocaine Group (Active Comparator): Lidocaine was administered through continuous infusion, immediately before induction of anesthesia
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2 mg/kg was administered through continuous infusion, immediately before induction of anesthesia
  Arms: Lidocaine Group
Drug: Magnesium Sulphate — Magnesium Sulphate 30 mg/kg was administered through continuous infusion, immediately before induction of anesthesia
  Arms: Magnesium Group

SUMMARY:
Justification and Objectives: The hemodynamic response to stimuli of the airways is a common phenomenon and its control is important to decrease systemic repercussions. The objective of this study is to compare the effects of intravenous administration of Magnesium Sulphate versus Lidocaine in the hemodynamics of this reflex after laryngoscopy and tracheal intubation. Methods: This double blind, randomized, single center, and prospective study evaluated 56 patients, ASA 1 or 2, aged between 18 and 65 years, scheduled for elective surgeries under general anesthesia with tracheal intubation. Patients were divided into two groups. Group M received 30mg/kg of Magnesium Sulphate, and group L 2 mg/kg of Lidocaine through continuous infusion, immediately before induction of anesthesia. The values for blood pressure (BP), heart rate (HR) and bispectral index (BIS) were measured in both groups at six distinct moments related to the administration of the drugs under study.

DETAILED DESCRIPTION:
This double-blind, randomized, single center, prospective study was approved by the Local Research Ethics Committee (FEPECS/SES-DF) under the report number 799.112 and has been identified on the Plataforma Brasil (http://aplicacao.saude.gov.br/plataformabrasil) under CAAE (Certificate of Presentation for Ethical Consideration) number 33365114.7.0000.5553. After written informed consent, 56 patients, ASA P1 or P2, aged between 18 and 65 years, scheduled for elective surgeries with orotracheal intubation (OTI), were assessed regarding their eligibility between the months of September and November, 2014 Of the 56 patients selected for the study according to the inclusion criteria, 7 were excluded during the evaluations, four from group M because of: frequent ventricular extrasystoles, introduction of nasal swab of adrenaline before the end of evaluations, intubation with video-laryngoscope and lack of sevoflurane in the vaporizer not checked during the evaluations. Three more patients were excluded from group L: one because of leakage of drugs (poorly secured venous access), another because of vomiting with consequent aspiration during ventilation with mask, and another for failed intubation in the first laryngoscopy.

When arriving in the surgery room, the patient was first identified, followed by standard monitoring with cardioscope (ECG), peripheral oxygen saturation (SpO2), noninvasive blood pressure (NIBP) and bispectral index (BIS). Venoclysis was performed at the discretion of the anesthesiologist, in accordance with the scale of the surgery/anesthesia ("Admission" time). Next, the pre-anesthetic medication was administered with midazolam (MDZ) in the dose of 0.05mg/kg. After two minutes (Time "2' after-MDZ"), the infusion with the drug under study was started, with a dose of 2mg/kg for lidocaine or 30mg/kg for magnesium sulphate, both diluted in 15mL of solution and infused in 10 minutes through a continuous infusion pump (CIP). After finishing the infusion (Time "End-CIP"), pre-oxygenation and anesthetic induction with intravenous fentanyl 2mcg/kg was performed, followed by propofol 2 mg/kg and rocuronium 0.6 mg/kg (Time "after-Ind"). The laryngoscopy was performed three minutes after the end of the rocuronium injection and if the BIS value was equal to or less than 50 (Time "after-OTI"). If the BIS value was not reached, a venous increment of 1mg/kg of propofol was administered. After orotracheal intubation, anesthesia was maintained through inhalation with sevoflurane 2%, and new measurements were taken after 3 and 6 minutes of intubation (Times "3' after-OTI" and "6' after-OTI"). Hypertension was considered when the BP values were 20% above baseline values or if Systolic Blood Pressure (SBP) > 140 mmHg. Hypotension was considered when the Blood Pressure (BP) values were 20% below baseline values or if SBP > 90 mmHg. Tachycardia was considered when the Heart Rate (HR) values were 20% above baseline values or if HR > 100 mmHg. Bradycardia was considered for HR values under 50 bpm.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2, aged between 18 and 65 years, scheduled for elective surgeries with orotracheal intubation at the Hospital de Base do Distrito Federal, Brazil

Exclusion Criteria:

* Patients who have contraindication or a history of hypersensitivity to the drugs involved in the work
* Patients with ischemic heart disease, atrioventricular block in any degree, diagnosed cardiac arrhythmias, heart failure
* Renal failure carrier
* Users of beta-blockers or calcium channel blockers,
* Patients who have forecast of difficult tracheal intubation,
* BMI < 35 kg/m2,
* Patients in whom neuroaxis block was performed before the induction of anesthesia,
* Patients who refused to participate in the study
* Those who needed two or more laryngoscopy attempts to position the orotracheal tube,
* Any other condition that, in the researchers' opinion, could offer risks to the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure Change in Systolic Blood Pressure | Within the first 6 minutes after oral intubation
  Qualification of hemodynamic response to oral intubation by the change in SBP after Magnesium Sulfate or Lidocaine infusion

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure | Within the first 6 minutes after oral intubation
  Qualification of hemodynamic response to oral intubation by the change in Diastolic Blood Pressure (DBP) after Magnesium Sulfate or Lidocaine infusion
Change in Heart Rate | Within the first 6 minutes after oral intubation
  Qualification of hemodynamic response to oral intubation by the change in HR after Magnesium Sulfate or Lidocaine infusion
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Within the first 6 minutes after oral intubation
  Hemodynamic stability analysis during anesthesia induction through the incidence of tachycardia, hypertension, bradycardia, hypotension and consumed vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, TSA, Principal Investigator — Hospital de Base do Distrito Federal, Brazil

REFERENCES:
- [Result] Nooraei N, Dehkordi ME, Radpay B, Teimoorian H, Mohajerani SA. Effects of intravenous magnesium sulfate and lidocaine on hemodynamic variables following direct laryngoscopy and intubation in elective surgery patients. Tanaffos. 2013;12(1):57-63. PMID 25191450